CLINICAL TRIAL: NCT03219749
Title: Examining the Effects of Exercise on Vascular Function in Obstructive Sleep Apnea
Brief Title: Sleep Apnea, Cardiovascular and Exercise Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Towson University (Other)
Collaborators: Pulmonary Critical Care Associates of Baltimore (Other)
Responsible Party: Principal Investigator, Devon Dobrosielski, Assistant Professor, Towson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R15HL133884 (NIH)
Record Dates: First submitted 2017-07-11; First posted 2017-07-17 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Obstructive Sleep Apnea; Vascular Diseases; Obesity
Keywords: obstructive sleep apnea; exercise training; vascular function
MeSH Terms: conditions — Sleep Apnea, Obstructive; Vascular Diseases; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Experimental): Exercise training will take place three times per week for six weeks and involve both aerobic and resistance exercise.
  Interventions: Behavioral: exercise training

INTERVENTIONS:
Behavioral: exercise training — Eligible participants will undergo 6 weeks of a combined aerobic and resistance exercise intervention. Training will take place 3 times per week for 1 hour. Forty minutes will be dedicated to aerobic training while 15 to 20 minutes will be devoted to resistance training.

SUMMARY:
Obstructive sleep apnea (OSA) results in vascular dysfunction, which increases the risk of cardiovascular disease. In contrast, exercise confers cardioprotection through improvements in vascular health. This proposal evaluates whether the beneficial effects of exercise on vascular function are attenuated in obese individuals suffering from untreated OSA.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a serious medical condition that affects an estimated 15 million US adults and is characterized by repeated episodes of upper airway obstruction, recurrent arousals and episodic oxyhemoglobin desaturations during sleep. These abnormalities contribute to subclinical alterations in vascular function that increase the risk of cardiovascular disease morbidity and mortality. In contrast, exercise decreases the risk of cardiovascular events and the promotion of physical activity continues to be at the top of our national public health agenda, as seen in the publication of the 1996 report of the US Surgeon General on physical activity and health. While the exact mechanisms for this protective benefit are not entirely clear, there is good evidence that exercise confers cardioprotection through its direct impact on vascular endothelial function. The American College of Sleep Medicine recommends exercise as a behavioral treatment option for OSA. Yet, most clinical trials upon which this recommendation is based have focused on establishing the effectiveness of lifestyle change (e.g., dietary induced weight loss and increased physical activity participation) for improving OSA severity in obese individuals, whereas less attention has been given to whether OSA moderates the effects of exercise on the cardiovascular disease substrate. The overarching hypothesis of this study is that OSA attenuates the beneficial effect of exercise on vascular function in obese individuals suffering from untreated OSA. The aims of the study are to 1) examine parameters of vascular function in obese persons with and without OSA, 2) evaluate the effects of an acute bout of exercise on brachial artery flow mediated dilation in obese persons with and without OSA, and 3) examine the effects of 6 weeks of exercise training on vascular function among those with and without OSA. These data will be immediately useful in clinical practice and inform how clinicians prescribe exercise and implement lifestyle changes to reduce cardiovascular disease risk in OSA patients.

ELIGIBILITY:
Inclusion Criteria:

- BMI between 30 and 42

Exclusion Criteria:

* Apnea-hypopnea index > 60 events (confirmed with overnight sleep study)
* Currently participating in an exercise program as defined as a minimum of moderate exercise > 30 minute/day, > 3 times or 90 minutes per week
* Participating in a weight loss program and NOT weight stable for 3 months
* History of heart disease
* Uncontrolled hypertension
* Cigarette smoking in the last 6 months
* Type 1 diabetes
* Women who are pregnant
* Currently using hormonal replacement therapy
* Comorbid conditions including concern, peripheral arterial disease, renal disease, lung disease, thyroid diseases, osteoporosis and arthritis with chronic joint pain

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in flow mediated dilation of the brachial artery | This outcome will be assessed at baseline and at 6 weeks
  Flow mediated dilation (in %) of the brachial artery will be assessed by vascular ultrasound

SECONDARY OUTCOMES:
exercise stress test | This outcome will be assessed at baseline and at 6 weeks
  The participant will walk on a treadmill. The treadmill speed and grade will continue to increase every 3 minutes until the participant can not continue due to fatigue. Physical fitness will be determined by measuring the amount of time the individual is able to continue on the treadmill before stopping.
dual energy X-ray absorptiometry | This outcome will be assessed at baseline and at 6 weeks
  The research participant lies on an examination table for approximately 10 minutes, during which time an X-ray type device scans the body and determines how much body mass is composed of fat tissue. This enables the investigator to monitor % body fat and determine if the exercise intervention influences body weight.
blood draw | This outcome will be assessed at baseline and at 6 weeks
  Markers of inflammation (e.g., C reactive protein, interleukin 6) will be assessed with chemical assays using a sample of blood drawn from the participant

CONTACTS AND LOCATIONS:
Locations (1):
- Towson University Wellness Center, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided